CLINICAL TRIAL: NCT00912548
Title: A Randomised Phase III Study for Evaluating the Role of the Addition of Ovarian Function Suppression to Tamoxifen in Young Women With Hormone-Sensitive Breast Cancer Who Remain in Premenopause or Regain Menstruation After Chemotherapy
Brief Title: Evaluating the Role of the Addition of Ovarian Function Suppression (OFS) to Tamoxifen in Young Women
Acronym: ASTRRA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Korean Breast Cancer Study Group (Other)
Responsible Party: Woo-Chul, Noh, Korea Cancer Center Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: KBCSG005
Record Dates: First submitted 2009-05-31; First posted 2009-06-03 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Breast Cancer
Keywords: premenopause; ovarian function suppression; tamoxifen
MeSH Terms: conditions — Breast Neoplasms | interventions — Goserelin; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- TAM+OFS(E) group (Experimental): Patients should be premenopausal women ,prior to the start of chemotherapy, less than or equal to 45 years of age with oestrogen receptor positive ± progesterone receptor positive who have undergone a primary mass excision, received an neo-/adjuvant chemotherapy ± radiotherapy for their stage I, II or III breast cancer. This arm is ovarian suppression group which have a various starting time of ovarian function suppression after neo-/adjuvant chemotherapy.
  Ovarian function suppression will be done by administration of LHRH agonist (ZOLADEXTM) for 2 years. After that, the patients will complete taking tamoxifen 20mg/day for 5 years.
  Interventions: Drug: goserelin; Drug: tamoxifen
- TAM(D) group (Active Comparator): Patients, less than or equal to 45 years of age with hormone receptor positive breast cancer will be enrolled. Included All the patients have already treated by surgery, neo- or adjuvant chemotherapy ±and/or radiotherapy before enrolment. At 0, 6, 12, 18 and 24 months since the baseline asTsessment(0), the ovarian function status will be evaluated by menstruation status or serum FSH level. If the patients are regarded as the premenopausal women, they will be randomized into the additional ovarian function suppression group or tamoxifen only group. The latter will complete taking tamoxifen 20mg/day for 5 years.
  Interventions: Drug: tamoxifen
- Permanent postmenopausal(A) group (No Intervention): Patients, less than or equal to 45 years of age with hormone receptor positive breast cancer will be enrolled. Included All the patients have already treated by surgery, neo- or adjuvant chemotherapy ±and/or radiotherapy before enrolment. Eligible patients except for premenopausal status at the baseline will be followed up until 2 years after the baseline assessment for evaluating the menopausal status. This group still remains to postmenopausal status and will taking tamoxifen 20mg/day for 5 years if they remain in the study.
- TAM(B) (Active Comparator): Patients, less than or equal to 45 years of age with hormone receptor positive breast cancer will be enrolled. Included All the patients have already treated by surgery, neo- or adjuvant chemotherapy ±and/or radiotherapy before enrolment. At 6, 12, 18 and 24 months since the baseline assessment (0), the ovarian function status will be evaluated by menstruation status or serum FSH level. If the patients are regarded as the premenopausal women, they will be randomized into the additional ovarian function suppression group or tamoxifen only group. This group, patients are premenopausal women, they will be randomized into tamoxifen only group, complete taking tamoxifen 20mg/day for 5 years.
  Interventions: Drug: tamoxifen
- TAM+OFS (C) (Experimental): Patients, less than or equal to 45 years of age with hormone receptor positive breast cancer will be enrolled. Included All the patients have already treated by surgery, neo- or adjuvant chemotherapy ±and/or radiotherapy before enrolment. At 6, 12, 18 and 24 months since the baseline assessment (0), the ovarian function status will be evaluated by menstruation status or serum FSH level. If the patients are regarded as the premenopausal women, they will be randomized. This group, patients are premenopausal women, they will be randomized into the additional ovarian function suppression group. Ovarian function suppression will be done by administration of LHRH agonist (ZOLADEXTM) for 2 years. Then, Patients will complete taking tamoxifen 20mg/day for 5 years.
  Interventions: Drug: goserelin; Drug: tamoxifen

INTERVENTIONS:
Drug: goserelin — 1. Zoladex™ administration:
     Zoladex™ depot is available as a sterile disposable syringe. The depot is administered subcutaneously under the abdominal skin under sterile conditions. If necessary the injection site may be pre-treated with a local anaesthetic.
  2. Sequence of administration Zoladex depot:
     The substance is administered for 24 months (2 years) at 28-day intervals (a period of 34 days between 2 administrations must not be exceeded).
  3. Dosage:
     Each depot contains 3.6mg Zoladex. The substance Zoladex is contained in a while cylindrical rodlet .
  4. Storage instructions for Zoladex™ Zoladex™ is kept a room temperature.
  Other Names: Zoladex®
  Arms: TAM+OFS (C); TAM+OFS(E) group
Drug: tamoxifen — 1. Dose and period of Tamoxifen therapy:
     Tamoxifen is administered in tablet form. Each day 2 X 10 mg or 1 X 20 mg Tamoxifen are taken in the form of the respective tablet.
  2. Storage instructions for Tamoxifen Tamoxifen is stored at room temperature away from light.
  Other Names: Nolvadex
  Arms: TAM(B); TAM(D) group; TAM+OFS (C); TAM+OFS(E) group

SUMMARY:
The purpose of this study is to compare 5-year disease free survival rate (DFS rate) between the hormone receptor positive breast cancer patients who were added Goserelin to Tamoxifen for ovarian function suppression after neo-/adjuvant cytotoxic chemotherapy and the hormone receptor positive breast cancer patients who were treated with Tamoxifen.

DETAILED DESCRIPTION:
* To compare overall Survival(OS) between the patients added Goserelin(ZOLADEXTM) to Tamoxifen and the patients treated with Tamoxifen alone in premenopausal status
* To compare 5-year disease free survival rate (DFS rate) between the patients who took tamoxifen only in postmenopause and the patients added Goserelin(ZOLADEXTM) to Tamoxifen for inducing ovarian function suppression in premenopause
* To determine the tolerability and safety of Tamoxifen with or without concomitant Zoladex

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have undergone excision of the primary breast mass, proven histologically to be invasive breast adenocarcinoma.
2. Patients must be within 3 months after the last cycle of chemotherapy.
3. Patients must have the history of normal menstruation prior to the start of chemotherapy.
4. Stage I, II or III
5. Woman, less than or equal to 45 years of age
6. Hormone receptor status : ER+ve and/or PgR+ve
7. WHO performance status 0, 1 or 2.
8. Patients who were treated with cytotoxic chemotherapy in pre- or post- surgery.
9. Adequate haematological function defined by haemoglobin 10g/dL, neutrophil count 1.5x109/L and platelets 100x109/L.
10. Adequate hepatic function defined by AST and ALT 2.5xupper limit of normal. Alkaline phosphatase 5xupper limit of normal, unless bone metastases in the absence of liver disease. Renal function adequate defined by creatinine<175mmol/L.

Exclusion Criteria:

1. Patients whose primary breast cancer was classified as:

   * ER(-),ER unknown
2. Patients with the history of hysterectomy or oophorectomy
3. Sarcomas or squamous cell carcinomas of the breast are not eligible.
4. Patients with malignancies (other than breast cancer) within the last 5 years, except for adequately treated in situ carcinoma of the cervix or basal cell / squamous cell carcinoma of the skin.
5. Investigational drugs given within the previous 4 weeks.
6. Patients known to be on any unlicensed non-cancer investigational agent.
7. Patients with thrombocytopaenia (platelets <100 x 109/l or on anti- coagulant therapy (contra-indicated due to risk of bleeding with i.m. injection of Zoladex).
8. Patients treated with CMF(cyclophosphamide/methotrexate/5-fluorouracil) as prior chemotherapy
9. Patients who are pregnant or lactating are ineligible.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1234 (Estimated)
Dates: Start 2009-05; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
all cause recurrence | the first 5 years after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Woo-Chul Noh, MD.PhD, Principal Investigator — Department of Surgery, Korea Cancer Center Hospital, 215-4 Gongneung-dong, Nowon-gu, Seoul, Korea
Locations (1):
- Department of Surgery, Korea Cancer Center Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim HJ, Noh WC, Nam SJ, Park BW, Lee ES, Im SA, Jung YS, Yoon JH, Kang SS, Park KH, Lee SJ, Jeong J, Lee MH, Cho SH, Kim SY, Kim HA, Han SH, Han W, Hur MH, Kim S, Ahn SH. Five-year changes in ovarian function restoration in premenopausal patients with breast cancer taking tamoxifen after chemotherapy: An ASTRRA study report. Eur J Cancer. 2021 Jul;151:190-200. doi: 10.1016/j.ejca.2021.03.017. Epub 2021 May 16. PMID 34010788
- [Derived] Kim HA, Lee JW, Nam SJ, Park BW, Im SA, Lee ES, Jung YS, Yoon JH, Kang SS, Lee SJ, Park KH, Jeong J, Cho SH, Kim SY, Kim LS, Moon BI, Lee MH, Kim TH, Park C, Jung SH, Gwak G, Kim J, Kang SH, Jin YW, Kim HJ, Han SH, Han W, Hur MH, Noh WC; Korean Breast Cancer Study Group. Adding Ovarian Suppression to Tamoxifen for Premenopausal Breast Cancer: A Randomized Phase III Trial. J Clin Oncol. 2020 Feb 10;38(5):434-443. doi: 10.1200/JCO.19.00126. Epub 2019 Sep 16. PMID 31518174
- [Derived] Kim HA, Ahn SH, Nam SJ, Park S, Ro J, Im SA, Jung YS, Yoon JH, Hur MH, Choi YJ, Lee SJ, Jeong J, Cho SH, Kim SY, Lee MH, Kim LS, Moon BI, Kim TH, Park C, Kim SJ, Jung SH, Park H, Gwak GH, Kang SH, Kim JG, Kim J, Choi SY, Lim CW, Kim D, Yoo Y, Song YJ, Kang YJ, Jung SS, Shin HJ, Lee KJ, Han SH, Lee ES, Han W, Kim HJ, Noh WC. The role of the addition of ovarian suppression to tamoxifen in young women with hormone-sensitive breast cancer who remain premenopausal or regain menstruation after chemotherapy (ASTRRA): study protocol for a randomized controlled trial and progress. BMC Cancer. 2016 May 19;16:319. doi: 10.1186/s12885-016-2354-6. PMID 27197523